CLINICAL TRIAL: NCT01522534
Title: Randomized Double Blind Controlled Trial Comparing a Blind Sciatic Nerve Block in the Popliteal Fossa to Intravenous Morphine for Traumatic Severe Acute Pain in the Prehospital Setting
Acronym: BPOP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough inclusions
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: chra-2009-001
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Injuries; Pain; Emergencies
Keywords: injuries; pain; Block, Nerve; morphine; Prehospital Emergency Care
MeSH Terms: conditions — Wounds and Injuries; Pain; Emergencies; Bites and Stings | interventions — Mepivacaine; Morphine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blind block with mepivacaine (Experimental): Blind block with mepivacaine and intravenous morphine
  Interventions: Drug: Mepivacaine
- Morphine (Active Comparator): Intravenous Morphine and placebo blind block
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Mepivacaine — mepivacaine 1% 20 ml corresponding to 200 mg
  Other Names: experimental group
  Arms: Blind block with mepivacaine
Drug: Morphine — Morphine alone with a placebo nerve block
  Other Names: control group
  Arms: Morphine

SUMMARY:
The purpose of the study is to determine the efficacity of a simple blind technic of loco regional anaesthesia of the sciatic nerve compared to the gold standard in emergency medecine : the intravenous morphine for treated the severe pain of leg, ankle or foot trauma in the prehospital setting and mountain rescue.

DETAILED DESCRIPTION:
Severe pain due to leg, ankle or foot trauma do not beneficiated of a simple loco regional anaesthesia technic. Loco regional anesthesia is superior to intravenous morphine for treating severe pain and specially during transportation and mobilization of the patient. The purpose of the study is to assessed a new technic of blind sciatic nerve block in the popliteal fossa in the pre hospital setting compared to the intravenous morphine. The blind technic is a modified technic of the classic sciatic nerve block with nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Severe pain (VAS > or = 60mm); injuries of the leg, ankle or foot

Exclusion Criteria:

* Hypersensitivity to student agents
* Local infection
* Nerve or vascular pathology in the affected limb, coagulation pathology,
* Chronic use of opoids, use of opoids within 6 hours
* Drug addiction
* Pregnancy
* Systolic blood pressure less than 90 mmHg
* Respiratory rate less than 16 per minute
* Glasgow coma scale < 14.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual analog scale pain score | 30 minutes

SECONDARY OUTCOMES:
Total dose of morphine | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Francois Xavier AGERON, MD, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (6):
- France (6):
  - Centre Hospitalier d'Albertville moutiers, Albertville
  - Centre Hospitalier de la Region d'Annecy, Annecy
  - Centre Hospitalier de Chambéry, Chambéry
  - Centre Hospitalier Universitaire de GRENOBLE, Grenoble
  - Centre medical d'Avoriaz, Morzine
  - Centre Hospitalier Sallanches Chamonix, Sallanches